CLINICAL TRIAL: NCT07181083
Title: Imaging-based Prediction of Stent-free Pharmaco-mechanical Thrombolysis in Patients With Extensive Acute Ilio-femoral Deep Vein Thrombosis
Brief Title: AI-Based Prediction Model for Iliofemoral DVT Thrombolysis
Status: Active, not recruiting | Type: Observational
Sponsor: Rajaie Cardiovascular Medical and Research Center (Other)
Responsible Party: Principal Investigator, Parham Sadeghipour, Doctor, Rajaie Cardiovascular Medical and Research Center
Other Study IDs: IR.RHC.REC.1403.013
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Deep Vein Thrombosis of the Lower Extremities
Keywords: Deep vein thrombosis; Prediction model; Iliofemoral vein; Pharmacomechanical thrombolysis; Magnetic resonance venography; Acute kidney injury
MeSH Terms: conditions — Venous Thrombosis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Extensive iliofemoral DVT: Patients with extensive ioliofemoral DVT candidate for pharmaco-mechanical thrombectomy
  Interventions: Device: Rheolytic thrombectomy

INTERVENTIONS:
Device: Rheolytic thrombectomy — Rheolytic thrombectomy via AngioJet ZelanteDVTTM Catheter (Boston Scientific Co., USA).

SUMMARY:
This prospective single-arm cohort study aims to develop an AI-powered prediction model for treatment outcomes in patients with acute extensive iliofemoral deep vein thrombosis (IF-DVT) undergoing stent-free pharmacomechanical thrombolysis. The study addresses the current lack of validated tools for patient selection and outcome prediction in catheter-directed interventions for proximal DVT.

Thirty consecutive adult patients with MRV-confirmed acute IF-DVT will undergo pharmacomechanical thrombolysis using the AngioJet ZelanteDVT system with adjunctive rtPA administration.

The primary objective is to develop a convolutional neural network (CNN) trained on serial MRV imaging data to predict three-month venous recanalization success. MRV acquisitions occur at baseline, predischarge, and three-month follow-up. Ground truth segmentation will be performed by an experienced radiologist using 3D Slicer, with semi-automated propagation across the dataset. Feature extraction will include geometric metrics, radiomic texture analysis, and morphological characteristics of both thrombus and vessel architecture.

Secondary endpoints include acute kidney injury incidence (a significant concern with rheolytic thrombectomy due to hemolysis-induced nephrotoxicity), post-thrombotic syndrome development assessed via Villalta scoring, and various safety outcomes including major bleeding per ISTH criteria.

The study protocol incorporates rigorous monitoring for AKI using KDIGO criteria, with systematic evaluation of renal function, hemolysis markers, and electrolyte balance. Hydration protocols and nephroprotective measures will be standardized, though specific strategies require clarification from the nephrology team.

This research addresses critical gaps in evidence-based patient selection for invasive DVT treatment, particularly following the mixed results of the ATTRACT trial. The AI prediction model could enable personalized treatment decisions, potentially improving the risk-benefit ratio of pharmacomechanical interventions while reducing unnecessary procedures in patients unlikely to benefit.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult (≥18 years) patients with an MRV-based diagnosis of acute IF- DVT
* Symptomatic patients with severe pain and\or leg swelling more than 5 cm
* Willing to participate in the study

Exclusion Criteria:

* Previous history of VTE
* Presence of DVT syndrome for more than 21 days
* Terminal systemic disease requiring palliative treatment
* Active bleeding
* History of hemorrhagic stroke
* Major fibrinolytic contraindication
* Any hereditary coagulopathy disorders
* Patients with baseline renal dysfunction with an estimated glomerular filtration rate (eGFR) of < 60 ml/min/1.73m2 due to Cockroft-Gault formula based on the creatinine level at the time of admission
* Having any underlying condition that makes the patient unsuitable for MRV and/or rheolytic thrombectomy procedure (e.g., allergy to contrast agent, claustrophobia)
* Having any underlying disabling condition that necessitates a prolonged complete bed rest prohibiting early ambulation
* Low-quality MRV imaging or motion artifact (exclusion criteria for the imaging sub-studies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be drawn from adult patients aged 18 years and older of both sexes presenting to the Rajaie Cardiovascular Medical and Research Institute, a tertiary referral cardiovascular center in Tehran, Iran, with acute symptomatic iliofemoral deep vein thrombosis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
During the procedure | 3 months post-procedure
  The extent of venous recanalization after stent-free pharmacomechanical thrombolysis as assessed by magnetic resonance venography at three months post-procedure. Recanalization will be graded as: Grade 0 (no flow/complete occlusion), Grade 1 (minimal flow with ≤25% lumen patency), Grade 2 (partial flow with 26-75% patency), or Grade 3 (near-complete flow with >75% patency). Treatment success is defined as achieving Grade 2 or 3 recanalization.

SECONDARY OUTCOMES:
MRV-based Predischarge Venous Recanalization | At hospital discharge (typically 3-7 days post-procedure)
  The extent of venous recanalization in the acute phase after stent-free pharmacomechanical thrombolysis as measured by magnetic resonance venography, classified as complete (>90% clearance), nearly complete (50-90% clearance), or partial (<50% resolution)
At hospital discharge (typically 3-7 days post-procedure) | 3 months post-procedure
  Quantified thrombus volume reduction from baseline to three-month follow-up as measured by magnetic resonance venography, with meaningful reduction defined as ≥50% volume decrease
MRV-based Predischarge Percentage Reduction in Thrombus Volume | At hospital discharge (typically 3-7 days post-procedure)
  Quantified thrombus volume reduction from baseline to hospital discharge as measured by magnetic resonance venography, with meaningful reduction defined as ≥50% volume decrease
Postprocedural Acute Kidney Injury Occurrence | During index hospitalization (typically 3-7 days)
  Development of acute kidney injury during hospitalization based on KDIGO criteria: ≥0.3 mg/dL increase in serum creatinine within 48 hours, ≥1.5x baseline creatinine increase, or urine output <0.5 mL/kg/h for 6 hours.
Need for New Renal Replacement Therapy | During index hospitalization (typically 3-7 days)
  Requirement for initiation of any form of renal replacement therapy (hemodialysis, continuous veno-venous hemofiltration, peritoneal dialysis) due to acute kidney injury in patients without previous dialysis history.
Postprocedural Oliguria or Anuria | During index hospitalization (typically 3-7 days)
  Development of oliguria (urine output <0.5 mL/kg/hour) or anuria (urine output <50 mL/day) during the index hospitalization period.
Postprocedural Hyperkalemia | During index hospitalization (typically 3-7 days)
  Elevated serum potassium concentration above normal limits (>5.0-5.5 mEq/L) during the index hospitalization period.
Postprocedural Gross Hematuria | During index hospitalization (typically 3-7 days)
  Presence of visible blood in urine detected by visual inspection or urine testing during the index hospitalization period.
Major Bleeding Events | During index hospitalization (typically 3-7 days)
  Major bleeding according to International Society of Thrombosis and Haemostasis (ISTH) definition: fatal bleeding, bleeding in critical organs, or bleeding causing ≥2.0 g/dL hemoglobin decrease or requiring ≥2 units red blood cell transfusion.
Three-month Recurrent Venous Thromboembolism | 3 months post-procedure
  Objectively confirmed recurrent symptomatic venous thromboembolism (deep vein thrombosis or pulmonary embolism) during the three-month follow-up period.
Three-month Post-thrombotic Syndrome Incidence | 3 months post-procedure
  Development of post-thrombotic syndrome defined as Villalta score ≥5, assessed through standardized evaluation of symptoms (pain, cramps, heaviness, paresthesia, pruritus) and clinical signs (edema, induration, hyperpigmentation, redness, venous ectasia, calf pain on compression).
Three-month Post-thrombotic Syndrome Severity | 3 months post-procedure
  Severity classification of post-thrombotic syndrome using Villalta score: mild (5-9), moderate (10-14), or severe (≥15 or venous ulceration).
In-hospital All-cause Mortality | During index hospitalization (typically 3-7 days)
  Death from any cause during the index hospitalization period.
Three-month All-cause Mortality | 3 months post-procedure
  Death from any cause during the three-month follow-up period.
Technical Success Rate | During the procedure
  Successful placement of the AngioJet device catheter and initiation of the thrombectomy procedure as intended per protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Rajaie Cardiovascular Medical and Research Institute, Tehran, Tehran Province, Iran